CLINICAL TRIAL: NCT02325791
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of a Human Monoclonal Antibody, REGN2222, for the Prevention of Medically Attended RSV Infection in Preterm Infants
Brief Title: Study to Evaluate the Efficacy and Safety of Suptavumab (REGN2222) for the Prevention of Medically Attended RSV (Respiratory Syncytial Virus) Infection in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R2222-RSV-1332
Record Dates: First submitted 2014-12-21; First posted 2014-12-25 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part A: Suptavumab 30 mg/kg (Experimental)
  Interventions: Drug: Suptavumab 30 mg/kg
- Part B: Placebo Matched to Suptavumab (Experimental)
  Interventions: Drug: Placebo Matched to Suptavumab
- Part B: Suptavumab 30 mg/kg- 1 Dose (Experimental)
  Interventions: Drug: Suptavumab 30 mg/kg- 1 Dose
- Part B: Suptavumab 30 mg/kg - 2 Doses (Experimental)
  Interventions: Drug: Suptavumab 30 mg/kg - 2 Doses

INTERVENTIONS:
Drug: Suptavumab 30 mg/kg — Participants received single dose of suptavumab 30 milligram per kilogram (mg/kg) intramuscularly (IM) on Day 1.
  Other Names: REGN2222
  Arms: Part A: Suptavumab 30 mg/kg
Drug: Placebo Matched to Suptavumab — Participants received 2 IM doses of placebo matched to suptavumab: the first dose on Day 1 and the second dose on Day 57.
  Arms: Part B: Placebo Matched to Suptavumab
Drug: Suptavumab 30 mg/kg- 1 Dose — Participants received single dose of suptavumab 30 mg/kg IM on Day 1 and single dose of placebo matched to suptavumab on Day 57.
  Arms: Part B: Suptavumab 30 mg/kg- 1 Dose
Drug: Suptavumab 30 mg/kg - 2 Doses — Participants received 2 doses of suptavumab 30 mg/kg IM: the first dose on Day 1 and the second dose on Day 57.
  Arms: Part B: Suptavumab 30 mg/kg - 2 Doses

SUMMARY:
The purpose of this study was to evaluate the efficacy, safety, pharmacokinetics (PK), and immunogenicity of suptavumab (REGN2222) in infants born no more than 35 weeks, 6 days gestational age who are no more than 6 months of age at the time of enrollment in their respective geographic location. In order to optimize the potential benefit in this vulnerable population, we conducted this study during the RSV season using dosing regimens that are expected to be effective.

DETAILED DESCRIPTION:
This study occurred in two parts: Part A and Part B.

Part A of the study was an open-label, PK evaluation of intramuscular (IM) administered suptavumab in preterm infants for whom palivizumab was not recommended to enable the selection of dosing regimens for Part B.

Part B of the study was randomized, double-blind, and placebo-controlled, designed to evaluate efficacy, safety, serum concentration and immunogenicity of IM administration of suptavumab in preterm infants for whom palivizumab was not recommended. The total duration of Part B was up to 265 days (includes a 28-day screening period, 57-day treatment period and 180-day follow-up period).

Up to 1515 subjects were planned to be included in Part B of the study. Participants were randomly assigned to 1 of 3 different groups, each with 505 infants; one group received one dose of suptavumab and one dose of placebo, the second group received two doses of suptavumab, and the third group received two doses of placebo.

There was a separate genetic testing sub study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Preterm, otherwise healthy male or female infant who is ≤6 months of age at the time of the first dose (i.e., infant must be treated on or before their 6 month birthday)
2. Gestational age is ≤35 weeks, 6 days at birth
3. Parent(s) or legal guardian(s) of the infant is able to understand the study requirements and willing to provide informed consent

Key Exclusion Criteria:

1. Eligible, recommended and have access to receive palivizumab per AAP or other local guidelines, standard practice, or by their healthcare provider
2. History of CLD defined as requirement of supplemental oxygen for 28 days after birth
3. Known hemodynamically significant congenital heart disease
4. Known immunodeficiency, neuromuscular disease, or congenital abnormalities of the airway
5. Known renal or hepatic dysfunction
6. Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
7. Known or suspected impairment of immunological functions or autoimmune diseases
8. History of anaphylaxis
9. Previously received palivizumab or any other investigational RSV prophylaxis or vaccine product
10. Previous reaction to IV immunoglobulin, blood products or other foreign proteins, including vaccines and monoclonal antibodies

Note: Other inclusion and exclusion criteria apply

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1177 (Actual)
Dates: Start 2015-07-21; Primary Completion 2017-07-05 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (205):
- United States (107):
  - Regeneron Investigational Site, Birmingham, Alabama
  - Regeneron Study Site, Mobile, Alabama
  - Regeneron Study Site, Little Rock, Arkansas
  - Regeneron Study Site, Anaheim, California
  - Regeneron Study Site, Bell Gardens, California
  - Regeneron Study Site, Dinuba, California
  - Regeneron Study Site, Downey, California
  - Regeneron Study Site, Huntington Beach, California
  - Regeneron Study Site, La Puente, California
  - Regeneron Study Site, Los Angeles, California
  - Regeneron Study Site, Madera, California
  - Regeneron Study Site, Palmdale, California
  - Regeneron Study Site, Ventura, California
  - Regeneron Study Site, West Covina, California
  - Regeneron Study Site, Aurora, Colorado
  - Regeneron Study Site, Thornton, Colorado
  - Regeneron Study Site, Hartford, Connecticut
  - Regeneron Study Site, Boynton Beach, Florida
  - Regeneron Study Site, Gainesville, Florida
  - Regeneron Study Site, Jacksonville, Florida
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, Orlando, Florida
  - Regeneron Study Site, Pensacola, Florida
  - Regeneron Study Site, Tampa, Florida
  - Regeneron Study Site, Winter Park, Florida
  - Regeneron Study Site, Atlanta, Georgia
  - Regeneron Study Site, Columbus, Georgia
  - Regeneron Study Site, Dalton, Georgia
  - Regeneron Study Site, Meridian, Idaho
  - Regeneron Study Site, Nampa, Idaho
  - Regeneron Study Site, Peoria, Illinois
  - Regeneron Study Site, South Bend, Indiana
  - Regeneron Study Site, Hutchinson, Kansas
  - Regeneron Study Site, Topeka, Kansas
  - Regeneron Study Site, Bardstown, Kentucky
  - Regeneron Study Site, Louisville, Kentucky
  - Regeneron Study Site, Metairie, Louisiana
  - Regeneron Study Site, New Orleans, Louisiana
  - Regeneron Study Site, Shreveport, Louisiana
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Site, Silver Spring, Maryland
  - Regeneron Study Site, Fall River, Massachusetts
  - Regeneron Study Site, Woburn, Massachusetts
  - Regeneron Study Site, Stevensville, Michigan
  - Regeneron Study Site, Duluth, Minnesota
  - Regeneron Study Site, Minneapolis, Minnesota
  - Regeneron Study Site, Saint Paul, Minnesota
  - Regeneron Study Site, Jackson, Mississippi
  - Regeneron Study Site, Bridgeton, Missouri
  - Regeneron Study Site, Kansas City, Missouri
  - Regeneron Study Site, Lincoln, Nebraska
  - Regeneron Study Site, Norfolk, Nebraska
  - Regeneron Study Site, Omaha, Nebraska
  - Regeneron Study Site, Reno, Nevada
  - Regeneron Study Site, Lebanon, New Hampshire
  - Regeneron Study Site, Neptune City, New Jersey
  - Regeneron Study Site, New Brunswick, New Jersey
  - Regeneron Study Site, Brooklyn, New York
  - Regeneron Study Site, Mineola, New York
  - Regeneron Study Site, New Hyde Park, New York
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, Rochester, New York
  - Regeneron Study Site, Syracuse, New York
  - Regeneron Study Site, The Bronx, New York
  - Regeneron Study Site, Boone, North Carolina
  - Regeneron Study Site, Chapel Hill, North Carolina
  - Regeneron Study Site, Durham, North Carolina
  - Regeneron Study Site, Raleigh, North Carolina
  - Regeneron Study Site, Cincinnati, Ohio
  - Regeneron Study Site, Cleveland, Ohio
  - Regeneron Study Site, Columbus, Ohio
  - Regeneron Study Site, Dayton, Ohio
  - Regeneron Study Site, Fairfield, Ohio
  - Regeneron Study Site, Mayfield Heights, Ohio
  - Regeneron Study Site, Toledo, Ohio
  - Regeneron Study Site, Youngstown, Ohio
  - Regeneron Study Site, Oklahoma City, Oklahoma
  - Regeneron Study Site, Tulsa, Oklahoma
  - Regeneron Study Site, Gresham, Oregon
  - Regeneron Study Site, Allentown, Pennsylvania
  - Regeneron Study Site, Erie, Pennsylvania
  - Regeneron Study Site, Hermitage, Pennsylvania
  - Regeneron Study Site, Charleston, South Carolina
  - Regeneron Study Site, Cheraw, South Carolina
  - Regeneron Study Site, Greenville, South Carolina
  - Regeneron Study Site, North Charleston, South Carolina
  - Regeneron Study Site, Alcoa, Tennessee
  - Regeneron Study Site, Kingsport, Tennessee
  - Regeneron Study Site, Nashville, Tennessee
  - Regeneron Study Site, Austin, Texas
  - Regeneron Study Site, Fort Sam Houston, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, San Antonio, Texas
  - Regeneron Study Site, Layton, Utah
  - Regeneron Study Site, Roy, Utah
  - Regeneron Study Site, St. George, Utah
  - Regeneron Study Site, Syracuse, Utah
  - Regeneron Study Site, Charlottesville, Virginia
  - Regeneron Study Site, Midlothian, Virginia
  - Regeneron Study Site, Richmond, Virginia
  - Regeneron Study Site, Vienna, Virginia
  - Regeneron Study Site, Huntington, West Virginia
  - Regeneron Study Site, Kingwood, West Virginia
  - Regeneron Study Site, Morgantown, West Virginia
  - Regeneron Study Site, Madison, Wisconsin
  - Regeneron Study Site, Marshfield, Wisconsin
  - Regeneron Study Site, Milwaukee, Wisconsin
- Regeneron Study Site, Hobart, Tasmania, Australia
- Bulgaria (13):
  - Regeneron Study Site, Sofia, Sofia-Grad
  - Regeneron Study Site, Kazanlak, Stara Zagora
  - Regeneron Study Site, Blagoevgrad
  - Regeneron Study Site, Dobrich
  - Regeneron Study Site, Gabrovo
  - Regeneron Study Site, Lom
  - Regeneron Study Site, Montana
  - Regeneron Study Site, Pleven
  - Regeneron Study Site, Plovdiv
  - Regeneron Study Site, Rousse
  - Regeneron Study Site, Silistra
  - Regeneron Study Site, Sliven
  - Regeneron Study Site, Vidin
- Canada (3):
  - Regeneron Study Site, Calgary, Alberta
  - Regeneron Study Site, Halifax, Nova Scotia
  - Regeneron Study Site, Ottawa, Ontario
- Chile (6):
  - Regeneron Study Site, La Florida, Santiago Metropolitan
  - Regeneron Study Site, Providencia, Santiago Metropolitan
  - Regeneron Study Site, Puente Alto, Santiago Metropolitan
  - Regeneron Study Site, Recoleta, Santiago Metropolitan
  - Regeneron Study Site, San José, Santiago Metropolitan
  - Regeneron Study Site, San Ramón, Santiago Metropolitan
- Denmark (4):
  - Regeneron Study Site, Aalborg
  - Regeneron Study Site, Hjørring
  - Regeneron Study Site, Næstved
  - Regeneron Study Site, Viborg
- Finland (4):
  - Regeneron Study Site, Oulu, Oulun Iaani
  - Regeneron Study Site, Tampere, Oulun Iaani
  - Regeneron Study Site, Pori
  - Regeneron Study Site, Turku
- Germany (14):
  - Regeneron Study Site, Bochum
  - Regeneron Study Site, Bramsche
  - Regeneron Study Site, Bretten
  - Regeneron Study Site, Frankenthal
  - Regeneron Study Site, Freiburg im Breisgau
  - Regeneron Study Site, Hamburg
  - Regeneron Study Site, Herxheim
  - Regeneron Study Site, Leipzig
  - Regeneron Study Site, Mainz
  - Regeneron Study Site, Mannheim
  - Regeneron Study Site, Mönchengladbach
  - Regeneron Study Site, Munich
  - Regeneron Study Site, Sankt Augustin
  - Regeneron Study Site, Wanzleben
- Hungary (6):
  - Regeneron Study Site, Szeged, Csongrád megye
  - Regeneron Study Site, Budapest
  - Regeneron Study Site, Gyula
  - Regeneron Study Site, Nyíregyháza
  - Regeneron Study Site, Pécs
  - Regeneron Study Site, Veszprém
- Regeneron Study Site, Utrecht, Netherlands
- New Zealand (3):
  - Regeneron Study Site, Palmerston North, Manawatu-Wanganui
  - Regeneron Study Site, Auckland, North Island
  - Regeneron Study Site, Wellington
- Regeneron Study Site, Panama City, Panama
- Regeneron Study Site, San Juan, Puerto Rico
- South Africa (3):
  - Regeneron Study Site, Johannesburg, Gauteng
  - Regeneron Study Site, Pretoria, Gauteng
  - Regeneron Study Site, Ga-Rankuwa, North West
- Spain (8):
  - Regeneron Study Site, Esplugues de Llobregat, Barcelona
  - Regeneron Study Site, A Coruña
  - Regeneron Study Site, Granada
  - Regeneron Study Site, Madrid
  - Regeneron Study Site, Manises
  - Regeneron Study Site, Málaga
  - Regeneron Study Site, Santiago de Compostela
  - Regeneron Study Site, Seville
- Sweden (2):
  - Regeneron Study Site, Gothenburg
  - Regeneron Study Site, Uppsala
- Turkey (Türkiye) (4):
  - Regeneron Study Site, Ankara
  - Regeneron Study Site, Istanbul
  - Regeneron Study Site, Izmir
  - Regeneron Study Site, Kocaeli
- Ukraine (10):
  - Regeneron Study Site, Chernivtsi, Chernivtsi Oblast
  - Regeneron Study Site, Dnipropetrovsk, Dnipropetrovsk Oblast
  - Regeneron Study Site, Odesa, Odesa Oblast
  - Regeneron Study Site, Vinnytsia, Vinnytsia Oblast
  - Regeneron Study Site, Kharkiv
  - Regeneron Study Site, Kyiv
  - Regeneron Study Site, Poltava
  - Regeneron Study Site, Sumy
  - Regeneron Study Site, Ternopil
  - Regeneron Study Site, Zaporizhzhia
- United Kingdom (14):
  - Regeneron Study Site, Coventry, Birmingham
  - Regeneron Study Site, Southampton, Hampshire
  - Regeneron Study Site, Gillingham, Kent
  - Regeneron Study Site, London, London, City of
  - Regeneron Study Site, Oldham, Manchester
  - Regeneron Study Site, Stockport, Manchester
  - Regeneron Study Site, Belfast
  - Regeneron Study Site, Birmingham
  - Regeneron Study Site, Glasgow
  - Regeneron Study Site, Manchester
  - Regeneron Study Site, Poole
  - Regeneron Study Site, Reading
  - Regeneron Study Site, Sheffield
  - Regeneron Study Site, Stockton-on-Tees

REFERENCES:
- [Derived] Simoes EAF, Forleo-Neto E, Geba GP, Kamal M, Yang F, Cicirello H, Houghton MR, Rideman R, Zhao Q, Benvin SL, Hawes A, Fuller ED, Wloga E, Pizarro JMN, Munoz FM, Rush SA, McLellan JS, Lipsich L, Stahl N, Yancopoulos GD, Weinreich DM, Kyratsous CA, Sivapalasingam S. Suptavumab for the Prevention of Medically Attended Respiratory Syncytial Virus Infection in Preterm Infants. Clin Infect Dis. 2021 Dec 6;73(11):e4400-e4408. doi: 10.1093/cid/ciaa951. PMID 32897368

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts between 21-Jul-2015 and 26-Sep-2017. Part A of study was conducted at 6 sites in 3 countries and Part B was conducted at 175 sites in 18 countries. Only Part B of the study was conducted in Europe. A total of 23 participants were enrolled in Part A and a total of 1,154 participants were randomized in Part B.
Pre-assignment Details: In Part A, 27 participants were screened, of which 23 received study drug. In Part B, out of 1,154 participants, 1,149 received first dose of study drug. Of those, 1,051 continued and received second dose 8 weeks later. Participants were randomized in 1:1:1 ratio in Part B by gestational age category & region (North America/Rest of World).
Groups:
- Part A: Suptavumab 30 mg/kg: Participants received single dose of suptavumab 30 milligram per kilogram (mg/kg) intramuscularly (IM) on Day 1.
- Part B: Placebo Matched to Suptavumab: Participants received 2 IM doses of placebo matched to suptavumab: the first dose on Day 1 and the second dose on Day 57.
- Part B: Suptavumab 30 mg/kg- 1 Dose: Participants received single dose of suptavumab 30 mg/kg IM on Day 1 and single dose of placebo matched to suptavumab on Day 57.
- Part B: Suptavumab 30 mg/kg - 2 Doses: Participants received 2 doses of suptavumab 30 mg/kg IM: the first dose on Day 1 and the second dose on Day 57.
Period: Overall Study
Arm/Group | Part A: Suptavumab 30 mg/kg | Part B: Placebo Matched to Suptavumab | Part B: Suptavumab 30 mg/kg- 1 Dose | Part B: Suptavumab 30 mg/kg - 2 Doses
Started | 23 | 383 | 385 | 381
Completed | 23 | 358 | 360 | 355
Not Completed | 0 | 25 | 25 | 26
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Death | 0 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 15 | 14 | 9
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 8 | 16

BASELINE CHARACTERISTICS:
Groups:
- Part B: Suptavumab 30 mg/kg - 2 Doses: Participants received 2 doses of suptavumab 30 mg/kg IM:the first dose on Day 1 and the second dose on Day 57.
- Total: Total of all reporting groups
Arm/Group | Part A: Suptavumab 30 mg/kg | Part B: Placebo Matched to Suptavumab | Part B: Suptavumab 30 mg/kg- 1 Dose | Part B: Suptavumab 30 mg/kg - 2 Doses | Total
Number analyzed (Participants) | 23 | 383 | 385 | 381 | 1172
Age, Customized [Count of Participants; unit: Participants]
  <=31 weeks 6 days | 5 | 62 | 59 | 59 | 185
  >=32 weeks & <=35 weeks 6 days | 18 | 321 | 326 | 322 | 987
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 186 | 172 | 179 | 546
  Male | 14 | 197 | 213 | 202 | 626
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 80 | 81 | 75 | 239
  Not Hispanic or Latino | 20 | 297 | 300 | 302 | 919
  Unknown or Not Reported | 0 | 6 | 4 | 4 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 2
  Asian | 0 | 2 | 3 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2 | 4
  Black or African American | 0 | 32 | 34 | 35 | 101
  White | 19 | 338 | 334 | 326 | 1017
  Other | 2 | 7 | 9 | 11 | 29
  Unknown or Not Reported | 0 | 4 | 3 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Part A: Serum Concentration of Suptavumab Over Time
Description: Part A was primarily designed to determine the pharmacokinetics (PK) of suptavumab in infants to inform the dose regimen used in Part B of the study. The study protocol specified the process and criteria for assessment of the dose. The dose used in Part B was to remain the same as Part A if the PK data up to Day 57 demonstrated that the individual PK observations were consistent with model-predicted concentrations, following age and body weight corrections.
Time Frame: Day 1 through Day 150
Population: The PK analysis set included participants who received a single dose of suptavumab and had at least 1 measurable concentration of suptavumab in serum. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specific time point.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Part A: Suptavumab 30 mg/kg - 1 Dose: Participants received a single dose of suptavumab 30 milligrams per kilogram (mg/kg) intramuscularly (IM) on Day 1.
Arm/Group | Part A: Suptavumab 30 mg/kg - 1 Dose
Number analyzed (Participants) | 22
mg/L
  Day 2: number analyzed (Participants) | 3
  Day 2 | 280 (92.9)
  Day 8: number analyzed (Participants) | 3
  Day 8 | 177 (40.2)
  Day 15: number analyzed (Participants) | 3
  Day 15 | 145 (28.7)
  Day 22: number analyzed (Participants) | 3
  Day 22 | 128 (3.21)
  Day 29: number analyzed (Participants) | 3
  Day 29 | 110 (10.3)
  Day 57: number analyzed (Participants) | 3
  Day 57 | 70.9 (7.62)
  Day 85: number analyzed (Participants) | 5
  Day 85 | 60.4 (14.0)
  Day 150 | 15.9 (7.88)

2. Primary Outcome: Part B: Percentage of Participants With Medically Attended Respiratory Syncytial Virus (RSV) Infection (Hospitalization or Outpatient Visit With Lower Respiratory Tract Infection [LRTI]) Up to Day 150
Description: A medically attended RSV infection defined as an infant with positive RSV test by Reverse-transcriptase polymerase chain reaction (RT-PCR) with any of following events: Hospitalized (on basis of assessment of admitting physician) for RSV infection or outpatient visit (emergency room [ER], urgent care [UC], or pediatric clinic visits [for either a sick or well visit]) with RSV lower respiratory tract infection (LRTI). An RSV LRTI in an infant: RSV proven respiratory infection (i.e positive RSV RT-PCR test) with parent(s)/guardian(s) report of cough/difficulty breathing, & with 1 of following signs of LRTI, as assessed by healthcare provider: - lower chest wall in drawing -hypoxemia (peripheral capillary oxygen saturation <95% breathing room air) - Wheezing/crackles. The 150-day efficacy assessment period: first study drug intake through the Day 150 visit.
Time Frame: From first study drug administration up to Day 150
Population: Full analysis set (FAS) included all randomized participants who received any study drug and was analyzed according to treatment allocated by Interactive voice response system (IVRS)/ Interactive web response system (IWRS) at randomization (as randomized).
Measure: Number; unit: Percentage of participants
Arm/Group | Part B: Placebo Matched to Suptavumab | Part B: Suptavumab 30 mg/kg- 1 Dose | Part B: Suptavumab 30 mg/kg - 2 Doses
Number analyzed (Participants) | 383 | 385 | 381
Percentage of participants | 8.1 | 7.7 | 9.3
Statistical Analysis 1: Comparison: Part B: Placebo Matched to Suptavumab vs Part B: Suptavumab 30 mg/kg - 2 Doses; A hierarchical inferential approach was used to control Type-1 error at 0.05 for pairwise comparisons of each suptavumab dose regimen to placebo. Missing values were imputed to KM estimate from the placebo group. Randomization strata adjusted in CMH test include region (North America vs. Rest of World) & gestational age category (<= 31 weeks 6 days GA vs >= 32 weeks 0 days and <= 35 weeks 6 days GA). Threshold for significance at 0.05 level; Test type: Superiority; p = 0.5773, Cochran-Mantel-Haenszel; percentage treatment difference = 1.15, 95% CI 2-sided [-2.898 to 5.201]
Statistical Analysis 2: Comparison: Part B: Placebo Matched to Suptavumab vs Part B: Suptavumab 30 mg/kg- 1 Dose; A hierarchical inferential approach was used to control Type-1 error at 0.05 for pairwise comparisons of each Suptavumab dose regimen to placebo. Missing values were imputed to Kaplan-Meier (KM) estimate from the placebo group. Randomization strata adjusted in Cochran-Mantel-Haenszel (CMH) test include region (North America vs. Rest of World) & gestational age category (<= 31 weeks 6 days GA vs >= 32 weeks 0 days and <= 35 weeks 6 days GA). Threshold for significance at 0.05 level; Test type: Superiority; Cochran-Mantel-Haenszel — Analysis performed using CMH statistics with randomization stratum adjusted using Mantel-Haenzel (MH) method to assess pairwise treatment difference (i.e. absolute risk reduction of each suptavumab arm compared to placebo; percentage treatment difference = -0.44, 95% CI 2-sided [-4.318 to 3.438]

3. Secondary Outcome: Part A: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in participants, who received investigational medicinal product (IMP) was considered an adverse event (AE) without regard to possibility of causal relationship with this treatment. TEAEs: AEs that developed/worsened/became serious during on-treatment period (defined as time between the date of first study drug administration & date of end of study/last visit).Serious AE: Any untoward medical occurrence that resulted in any of following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious & non-serious AEs. National Cancer Institute Common Terminology Criteria (NCI-CTCAE) version 4.03(Grade 3 [severe] & Grade 4[life-threatening]) was used in this study to grade clinical AEs.
Time Frame: Baseline through Day 150
Population: Safety analysis set (SAF) included participants who received any dose of suptavumab.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Suptavumab 30 mg/kg
Number analyzed (Participants) | 23
Percentage of participants
  Any TEAE | 69.6
  Any Grade 3/Serious TEAE | 4.3

4. Secondary Outcome: Part B: Serum Concentration of Suptavumab
Description: Serum samples for drug concentration will be collected at pre-specified time points
Time Frame: Day 29, 57, 85, 113 and Day 150 Post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligram per liter (mg/L)
Arm/Group | Part B: Suptavumab 30 mg/kg- 1 Dose | Part B: Suptavumab 30 mg/kg - 2 Doses
Number analyzed (Participants) | 386 | 334
Milligram per liter (mg/L)
  Day 29: number analyzed (Participants) | 11 | 14
  Day 29 | 142 (45.5) | 145 (43.4)
  Day 57: number analyzed (Participants) | 62 | 55
  Day 57 | 95.6 (44.2) | 93.5 (29.8)
  Day 85: number analyzed (Participants) | 96 | 85
  Day 85 | 70.1 (29.0) | 238 (52.9)
  Day 113: number analyzed (Participants) | 96 | 94
  Day 113 | 38.1 (20.1) | 149 (54.0)
  Day 150: number analyzed (Participants) | 359 | 314
  Day 150 | 18.7 (9.89) | 70.6 (26.4)

5. Secondary Outcome: Part B: Number of Participants With At Least One Positive Anti-Drug Antibody (ADA) Assay
Description: ADA category of each participant was classified as pre-existing immunoreactivity (a positive ADA response at baseline with a <4-fold increase in titer for all post baseline samples), treatment-boosted (a positive response at baseline with at least one post baseline titer at >=4-fold the baseline titer), or treatment-emergent (TE [any positive post baseline assay response when baseline results were negative or missing]). TE ADA responses were further classified as persistent (treatment-emergent positive ADA response detected in at least 2 consecutive post baseline samples separated by at least a 12-week post baseline period [based on nominal sampling time], with no ADA-negative samples in-between, regardless of any missing samples or a positive response at the last ADA sampling time point), indeterminate (a positive assay response at the last collection time point only, regardless of any missing samples), or transient (not persistent/indeterminate, regardless of any missing samples).
Time Frame: Day 1 through Day 150
Population: The ADA analysis set contained participants who received a single dose of suptavumab and had at least 1 post-treatment ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo Matched to Suptavumab | Part B: Suptavumab 30 mg/kg- 1 Dose | Part B: Suptavumab 30 mg/kg - 2 Doses
Number analyzed (Participants) | 363 | 389 | 336
Participants
  Negative/Pre-Existing | 351 | 380 | 336
  Treatment Boosted | 0 | 0 | 0
  Treatment-Emergent | 12 | 9 | 0
  Treatment-Emergent: Persistent | 0 | 0 | 0
  Treatment-Emergent: Transient | 1 | 0 | 0
  Treatment-Emergent: Indeterminate | 11 | 9 | 0

6. Secondary Outcome: Part B: Percentage of Participants Hospitalized With Medically Attended RSV Infection or Outpatient Visit Lower Respiratory Tract Infection (LRTI) or Upper Respiratory Tract Infection (URTI) Up to Day 150
Description: A medically attended RSV infection was defined as an infant with a positive RSV test by RT-PCR with any of the following events: -Hospitalized (on the basis of the assessment of the admitting physician) for RSV infection - or Outpatient visit (ER, UC), or pediatric clinic visits [for either a sick or well visit]) with RSV LRTI. An RSV LRTI in an infant: RSV-proven respiratory infection (i.e, positive RSV RT-PCR test) with parent(s)/guardian(s) report of cough or difficulty breathing, and with 1 of the following signs of LRTI, as assessed by a healthcare provider: -Lower chest wall indrawing -Hypoxemia (peripheral capillary oxygen saturation <95% breathing room air) -Wheezing or crackles. The 150-day efficacy assessment period:first study drug intake through the Day 150 visit.
Time Frame: From the first study drug administration up to Day 150
Population: Analysis was performed on FAS population.
Measure: Number; unit: Percentage of participants
Arm/Group | Part B: Placebo Matched to Suptavumab | Part B: Suptavumab 30 mg/kg- 1 Dose | Part B: Suptavumab 30 mg/kg - 2 Doses
Number analyzed (Participants) | 383 | 385 | 381
Percentage of participants | 12.5 | 11.9 | 14.5
Statistical Analysis 1: Comparison: Part B: Placebo Matched to Suptavumab vs Part B: Suptavumab 30 mg/kg- 1 Dose; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Cochran-Mantel-Haenszel; percentage treatment difference = -0.67, 95% CI 2-sided [-5.291 to 3.959]
Statistical Analysis 2: Comparison: Part B: Placebo Matched to Suptavumab vs Part B: Suptavumab 30 mg/kg - 2 Doses; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Cochran-Mantel-Haenszel; percentage treatment difference = 2.02, 95% CI 2-sided [-2.836 to 6.867]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Part A: Day 150 and Part B: Day 237) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are TEAEs that developed/worsened during the 'on treatment period'. On treatment period for Part A: Day from first dose of drug to the End of study i.e. Day 150 & for Part B: Day from first dose of drug up to the day of last dose of drug plus 180 days. Safety analysis set. Participant data was summarized according to treatment group.
Groups:
- Part A: Suptavumab 30 mg/kg: Participants received single dose of suptavumab 30 mg/kg IM on Day 1.
Arm/Group | Part A: Suptavumab 30 mg/kg | Part B: Placebo Matched to Suptavumab | Part B: Suptavumab 30 mg/kg- 1 Dose | Part B: Suptavumab 30 mg/kg - 2 Doses
All-Cause Mortality (participants affected / at risk) | 0/23 | 3/384 | 1/418 | 0/348
Serious Adverse Events (participants affected / at risk) | 0/23 | 44/384 | 54/418 | 29/348
Other Adverse Events (participants affected / at risk) | 13/23 | 218/384 | 219/418 | 198/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Suptavumab 30 mg/kg (N=23) | Part B: Placebo Matched to Suptavumab (N=384) | Part B: Suptavumab 30 mg/kg- 1 Dose (N=418) | Part B: Suptavumab 30 mg/kg - 2 Doses (N=348)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-Respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Amniotic band syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macrocephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Sandifer's syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crying (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 9 (9) | 10 (11) | 7 (7)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pseudocroup (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 5 (6) | 13 (13) | 2 (2)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 5 (5) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respirovirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Eye haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-Abdominal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotonic-Hyporesponsive episode (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Apnoea neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Child abuse (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Suptavumab 30 mg/kg (N=23) | Part B: Placebo Matched to Suptavumab (N=384) | Part B: Suptavumab 30 mg/kg- 1 Dose (N=418) | Part B: Suptavumab 30 mg/kg - 2 Doses (N=348)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 13 (13) | 16 (16) | 11 (11)
Constipation (Gastrointestinal disorders) | 0 (0) | 20 (20) | 11 (13) | 14 (14)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 15 (16) | 24 (25) | 12 (13)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 31 (32) | 25 (25) | 24 (26)
Pyrexia (General disorders) | 0 (0) | 31 (40) | 32 (37) | 22 (24)
Bronchiolitis (Infections and infestations) | 2 (2) | 16 (19) | 19 (27) | 27 (33)
Bronchitis (Infections and infestations) | 0 (0) | 24 (32) | 24 (30) | 13 (20)
Conjunctivitis (Infections and infestations) | 1 (1) | 18 (20) | 25 (28) | 18 (20)
Nasopharyngitis (Infections and infestations) | 0 (0) | 53 (73) | 30 (35) | 35 (45)
Otitis media (Infections and infestations) | 0 (0) | 29 (41) | 49 (84) | 26 (37)
Rhinitis (Infections and infestations) | 1 (1) | 14 (15) | 17 (18) | 18 (19)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 74 (102) | 92 (127) | 75 (119)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 20 (26) | 19 (26) | 21 (24)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 14 (20) | 24 (27) | 23 (24)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 25 (35) | 24 (27) | 27 (33)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 12 (13) | 8 (8) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (3):
  • Study Protocol (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT02325791/Prot_000.pdf
  • Statistical Analysis Plan: Part A (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT02325791/SAP_001.pdf
  • Statistical Analysis Plan: Part B (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT02325791/SAP_002.pdf